CLINICAL TRIAL: NCT06191185
Title: IMProving Adherence to Colonoscopy Through Teams and Technology
Acronym: IMPACTT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Diagnostic
Other Study IDs: P0555149; R01CA271031 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer; Cancer Colorectal; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Best Practices Bundle (BPB), No Patient Instructions and Navigation (PIN) (Experimental): BPB: patient tracking and lists, audit and feedback, standardized documentation, standardization of care team communication.
  No PIN: Patients will receive usual communication from their care team.
  Interventions: Behavioral: BPB, No PIN
- BPB, PIN (Experimental): BPB: patient tracking and lists, audit and feedback, standardized documentation, standardization of care team communication.
  PIN: enhanced patient instructions and navigation (PIN).
  Interventions: Behavioral: BPB, PIN
- No BPB, PIN (Experimental): No BPB: Clinic's usual practice after a patient receives an abnormal FIT result.
  PIN: enhanced patient instructions and navigation (PIN).
  Interventions: Behavioral: No BPB, PIN
- No BPB, No PIN (Experimental): No BPB: Clinic's usual practice after a patient receives an abnormal FIT result.
  No PIN: Patients will receive usual communication from their care team.
  Interventions: Behavioral: No BPB, No PIN

INTERVENTIONS:
Behavioral: BPB, No PIN — Patient-level: standard communication from care team.
  Clinic-level: A program of "best practices" will be implemented to improve team communication, optimize practice workflow, and identify and track patients with abnormal FIT results through colonoscopy completion.
  Arms: Best Practices Bundle (BPB), No Patient Instructions and Navigation (PIN)
Behavioral: BPB, PIN — Patient-level: The patient-facing evidence-based instructions, communication, and navigation part of the intervention will leverage the short messaging service (SMS) text messaging platform, HealthySMS.
  Clinic-level: A program of "best practices" will be implemented to improve team communication, optimize practice workflow, and identify and track patients with abnormal FIT results through colonoscopy completion.
  Arms: BPB, PIN
Behavioral: No BPB, PIN — Patient-level: The patient-facing evidence-based instructions, communication, and navigation part of the intervention will leverage the SMS text messaging platform, HealthySMS.
  Arms: No BPB, PIN
Behavioral: No BPB, No PIN — Patient-level: standard communication from their care team.
  Arms: No BPB, No PIN

SUMMARY:
Complete and timely colonoscopy after an abnormal stool-based colorectal cancer screening test results in early detection, cancer prevention, and reduction in mortality, but follow-up in safety-net health systems occurs in less than 50% at 6 months. The proposal will implement multi-level approach consisting of a stepped-wedge clinic-level intervention of team-based best practices co-developed with primary and specialty care, a patient-level technology intervention to provide enhanced instructions and navigation to complete diagnostic colonoscopy, and a mixed methods evaluation to explore multi-level factors contributing to intervention outcomes. Developing a solution to this high-risk and diverse population has the potential to translate to other health systems, support patient self-management, and address other patient conditions.

DETAILED DESCRIPTION:
Follow-up colonoscopy after abnormal stool-based colorectal cancer screening (e.g., fecal immunochemical test (FIT)) results in early detection of colorectal cancer (CRC), prevention of CRC, and reduction in CRC mortality. FIT is a commonly utilized screening test that can be performed at home, is inexpensive, scalable, and often adopted in health systems where colonoscopy resources are scarce. Despite evidence that timely colonoscopy is necessary after an abnormal FIT result, completion of colonoscopy occurs in less than 50% of patients at 6 months and varies significantly by clinic and health systems. In addition to understanding the meaning of an abnormal FIT, three care transitions must occur smoothly for the patient: colonoscopy referral, scheduling, and attendance. However, multilevel factors influence missed follow-up, and multilevel solutions are needed along the care continuum to address clinic-, provider-, and patient-level factors that impair or delay colonoscopy completion.

IMProving Adherence to Colonoscopy through Teams and Technology (IMPACTT), proposes to close gaps and reduce disparities in CRC screening by improving the completion of diagnostic colonoscopy following abnormal FIT in vulnerable populations using a multilevel approach consisting of interventions at the clinic-, provider- and patient-level. The specific aims are 1) to evaluate the effect of a clinic-level intervention targeting primary care providers and staff to adopt "best practices" to support colonoscopy completion in patients with abnormal FIT results, 2) to determine the effect of a patient-level technology intervention with enhanced instructions and navigation for patients with abnormal FIT to complete a diagnostic colonoscopy, and 3) to explore the multilevel implementation factors contributing to intervention outcomes using mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abnormal FIT result
* Patients ages 18 years or older
* English, Spanish, or Cantonese speaking

Exclusion Criteria:

* Patients with normal FIT result
* Patients younger than age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Colonoscopy completion | 6 months after abnormal FIT result
  Wait time for routine colonoscopy is often less than 6 weeks and less than 2 weeks if one is willing to take an afternoon appointment. Completion of colonoscopy will be captured by extracting pertinent colonoscopy elements

SECONDARY OUTCOMES:
Quality of bowel preparation | At time of colonoscopy procedure
  The quality of procedure preparation is defined as excellent, good, fair, and poor.
Referred to GI for colonoscopy | 6 weeks after abnormal FIT result
  After an abnormal FIT result, providers should review the test result, communicate with patients, and refer the patient to GI to complete a colonoscopy.
Scheduled by GI for colonoscopy | 8 weeks after GI referral
  After an abnormal FIT result, providers will refer patients. The electronic referral is reviewed by GI, who will call the patient to schedule the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Urmimala Sarkar, MD, MPH, Principal Investigator — University of California, San Francisco; Ma Somsouk, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Wong J, Avilez L, Olazo K, Olanrewaju S, McCulloch CE, Pasick R, Patel S, Somsouk M, Sarkar U. Multilevel intervention for follow-up of abnormal FIT in the safety-net: IMProving Adherence to Colonoscopy through Teams and Technology (IMPACTT). Contemp Clin Trials. 2025 Mar;150:107810. doi: 10.1016/j.cct.2025.107810. Epub 2025 Jan 12. PMID 39809342